CLINICAL TRIAL: NCT03790696
Title: A Novel Mechanism-Based Treatment for Pediatric Anxiety Disorders
Brief Title: Novel Anxiety Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201702012
Record Dates: First submitted 2018-12-18; First posted 2019-01-02 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Cognitive Training; Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study is a randomized control trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomized to active vs. sham treatment on a 50/50 basis. The participants and the staff performing the pre- and post- treatment psychiatric interviews will remain blinded throughout the study. Study staff administering the treatment will be aware of the active vs. sham status of the participant, in order to deliver and monitor the appropriate cognitive training program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Cognitive Training (Experimental): Participants will complete 30-45 minute cognitive training program twice a week for four weeks.
  Interventions: Device: Cognitive Training Program
- Sham Cognitive Training (Sham Comparator): Participants will complete 30-45 minute cognitive training program twice a week for four weeks.
  Interventions: Device: Cognitive Training Program

INTERVENTIONS:
Device: Cognitive Training Program — The cognitive training program has been designed by Dr. Sylvester. It is a simple computer game looking at some shapes and faces on a computer screen and pressing a button when a target shape appears.
  This is the first study to use this exact computer training regimen for testing in its ability to reduce symptoms of anxiety in children with anxiety disorders. Each session of the computer game takes approximately 45-60 minutes and subjects complete 8 total sessions over one month. The computer game involves paying attention to parts of the screen while distracting square boxes appear at other locations. A target "X" appears at the location that participants are paying attention to and the subjects press a button when it appears.
  Other Names: novel computer-based cognitive training program; computer-delivered cognitive training program

SUMMARY:
The first aim of this study, as mentioned in the attached NIH grant, is to test the feasibility and acceptability of a novel computer-based cognitive training program that is designed to rehabilitate the brain's ventral attention network (VAN), a brain system associated with anxiety disorders.

Once feasibility and acceptability is determined the investigators will begin aim 2 where the investigators will test the efficacy of this novel treatment, which could reduce the symptoms of anxiety disorders in children (and adults) by training them to actively ignore stimuli in turn reducing the activity of the VAN. To test this potential treatment the investigators will recruit 60 children with anxiety disorders and 10 healthy children to compare an active version of a computer training program to a sham version of training. The investigators will also measure VAN reactivity before and after treatment using functional magnetic resonance imaging (fMRI). The rationale of this research is that it could lead to a novel, safe, mechanism-based treatment for a major public health problem.

DETAILED DESCRIPTION:
Children will be recruited through local schools, pediatricians' offices, and through Dr. Sylvester's child anxiety clinic by asking staff to present Institutional Review Board (IRB) approved recruitment materials to potentially interested families. The investigators will also recruit with advertisements and placement of approved flyers, paragraphs and materials throughout the greater Washington University community as well as throughout the St. Louis community.

The research assistant will make 'screening materials' available to recruitment sites including schools and pediatricians' offices. Staff at these recruitment sites will identify potential participants and distribute materials accordingly. Staff will only provide recruitment materials and will not answer questions regarding the study -- all questions will be answered by study staff. Screening materials will include a consent script, the contact information sheet, the SCARED, and the MFQ.

A member of the research team will review screening materials and contact potential participants by phone on the basis of meeting inclusion criteria. This member of the research team will provide parent participants with information about the study and required elements of consent over the telephone (see attached "Initial Phone Screen") prior to obtaining the parent's verbal consent to participate in the screening elements of the study (Initial Phone Screen as well as SCARED/MFQ).

If a parent and child meet eligibility criteria for enrollment in the study based on their Initial Phone Screen, and parents indicate they wish to continue with the study, the research team will arrange an in-person assessment. On the day of the in-person assessment, a research assistant will provide ample time for the parents to read/review the consent form and will answer any questions the parent may have prior to signing. Research team members will remind participants that their participation is completely voluntary and they can choose to withdraw at any time.

After the in-person assessment, the participant may be asked to return for another visit to complete functional magnetic resonance imaging. This additional visit will be optional and not a requirement of participation in the overall study. The subject can choose not to participate in this phase of the study and may withdraw at any time. If the subject is interested, the investigators will obtain a separate document of informed consent for the imaging phase. As in the original informed consent document, immediately after the in-person assessment, a research assistant will provide ample time for the parents to read/review the imaging consent form and will answer any questions the parent may have prior to signing.

The research assistant may also ask the participants at the end of the in-person assessment whether the investigators could call them in the future to participate in the imaging phase of the study. If the participant agrees, the team will call the participant within the next 3 months to set up an appointment. In this case, the informed consent for imaging would be obtained at the beginning of the imaging visit with all of the above procedures applying.

ELIGIBILITY:
Inclusion Criteria:

* ages of 8-12
* have a current diagnosis of separation anxiety disorder, generalized anxiety disorder, and/or social phobia.

Exclusion Criteria:

* prior diagnoses of attention deficit hyperactivity disorder (ADHD)
* autism spectrum disorder
* intellectual disability (IQ<70)
* a significant medical problem
* current use of psychotropic medication other than selective serotonin reuptake inhibitor (SSRI) (children who are currently taking an SSRI and are still experiencing symptoms of anxiety will not be excluded).

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washinton University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the Novel Anxiety Treatment Study took place from 2/2/2017 until 12/20/2019. Recruitment was primarily done at pediatrician offices and elementary schools in the St. Louis Metropolitan area. Recruitment ended early due to COVID-19.
Pre-assignment Details: Several participants met eligibility criteria for the study, but ultimately did not participate due to withdrawing prior to baseline (2), issues with the time commitment required (1), or not responding to research staff/not being scheduled (4).
  Overall we consented 21 child/parent dyads. 2 dyads were excluded after baseline due to no clinical anxiety present and 1 dyad was excluded due to the COVID pandemic starting. 18 child/parent dyads were assigned a training program.
Groups:
- Active Cognitive Training: Participants will complete 30-45 minute cognitive training program twice a week for four weeks.
  Cognitive Training Program: The cognitive training program has been designed by Dr. Sylvester. It is a simple computer game looking at some shapes and faces on a computer screen and pressing a button when a target shape appears.
  This is the first study to use this exact computer training regimen for testing in its ability to reduce symptoms of anxiety in children with anxiety disorders. Each session of the computer game takes approximately 45-60 minutes and subjects complete 8 total sessions over one month. The computer game involves paying attention to parts of the screen while distracting square boxes appear at other locations. A target "X" appears at the location that participants are paying attention to and the subjects press a button when it appears.
- Sham Cognitive Training: Participants will complete 30-45 minute cognitive training program twice a week for four weeks.
  Cognitive Training Program: The cognitive training program has been designed by Dr. Sylvester. It is a simple computer game looking at a fixation cross and pressing a button when a target shape appears.
  This is the first study to use this exact computer training regimen for testing in its ability to reduce symptoms of anxiety in children with anxiety disorders. Each session of the computer game takes approximately 45-60 minutes and subjects complete 8 total sessions over one month. The computer game involves paying attention to parts of the screen and in the sham training, there are no distractor boxes. A target "X" appears at the location that participants are paying attention to and the subjects press a button when it appears.
Period: Overall Study
Arm/Group | Active Cognitive Training | Sham Cognitive Training
Started | 10 (Parent/child dyads were consented to the study but only child completed cognitive training - 10 children were assigned to the active cognitive training and each of these children had a parent (10 parents total) who consented to participate in the study (interviews/surveys)) | 8 (8 children were assigned to the sham cognitive training and each of these children had a parent (8 parents total) who consented to participate in the study (interviews/surveys))
Completed | 10 (10 children completed the active cognitive training, and each of these children had a parent (10 parents total) who completed their portion of the research study (interview/surveys)) | 7 (7 children completed the sham cognitive training and each of these children had a parent (7 parents total) who completed their portion of the research study (interview/surveys))
Not Completed | 0 | 1
Not completed — Cognitive training task was too difficult for child to complete. | 0 | 1

BASELINE CHARACTERISTICS:
Population: Child participants were randomized after completing the baseline assessment and still meeting eligibility criteria for the study. Parents of the children reported on their child at the baseline and post treatment assessments. Baseline Characteristics data were not collected for parents.
Groups:
- Sham Cognitive Training: Participants will complete 30-45 minute cognitive training program twice a week for four weeks.
  Cognitive Training Program: The cognitive training program has been designed by Dr. Sylvester. It is a simple computer game looking at some shapes and faces on a computer screen and pressing a button when a target shape appears.
  This is the first study to use this exact computer training regimen for testing in its ability to reduce symptoms of anxiety in children with anxiety disorders. Each session of the computer game takes approximately 45-60 minutes and subjects complete 8 total sessions over one month. The computer game involves paying attention to parts of the screen, no distractor boxes appear in the sham training. A target "X" appears at the location that participants are paying attention to and the subjects press a button when it appears.
- Total: Total of all reporting groups
Arm/Group | Active Cognitive Training | Sham Cognitive Training | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 8 | 18
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.82 (1.17) | 11.09 (1.75) | 10.36 (1.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 9 | 7 | 16
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Symptoms of Anxiety Based on Screen for Anxiety and Related Disorders (SCARED) Parent Report at Baseline and Post Assessment
Description: Another outcome will be change in symptoms of anxiety as measured by the SCARED at the baseline and post training assessments. These scores will be subtracted (post training assessment - baseline assessment) to see the change in anxiety symptoms from the beginning of the study to post treatment. A total score of >25 may indicate the presence of an Anxiety Disorder. Scores higher than 40 are more specific based on the total score for specific items. Scores for the SCARED can range from 0-82.
Time Frame: Children/Caregivers will complete the SCARED measure at their baseline appointment before beginning treatment as well as at their final appointment after 4 weeks of completing the training.
Population: This population was recruited through pediatrician offices and elementary schools. All children met DSM-5 criteria for GAD, Social Phobia, or Separation Anxiety Disorder.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Active Training Participants: Participants who completed the active cognition training
- Sham Training Participants: Participants who completed the sham cognitive training
Arm/Group | Active Training Participants | Sham Training Participants
Number analyzed (Participants) | 10 | 8
units on a scale | -20.4 [-30.17 to -10.63] | -21.12 [-24.93 to -17.32]

2. Secondary Outcome: Change in Symptoms of Anxiety Based on Screen for Anxiety and Related Disorders (SCARED) Child Report at Baseline and Post Assessment
Description: as for outcome 1
Time Frame: as for outcome 1
Population: This population was recruited through pediatrician offices and elementary schools. All children met DSM-5 criteria for GAD, Social Phobia, or Separation Anxiety Disorder. We looked at improvement in anxiety across all participants (both active and sham training) since our dataset was smaller than anticipated.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Active Training Participants: change in anxiety for active training participants
- Sham Training Participants: change in anxiety for sham training participants
Arm/Group | Active Training Participants | Sham Training Participants
Number analyzed (Participants) | 10 | 8
units on a scale | -11.3 [-20.48 to -2.13] | -9.75 [-17.32 to -2.18]

3. Secondary Outcome: Change in Symptoms of Anxiety Based on Pediatric Anxiety Rating Scale (PARS) From Baseline to Post Assessment.
Description: Secondary outcomes will include the change in symptoms of anxiety on the PARS and diagnostic status. The investigators will test whether active versus sham training significantly changes symptoms in children with anxiety disorders. This will be calculated by subtracting (PARS post treatment - PARS before treatment)
  The PARS is a clinician-administered measure of pediatric anxiety that incorporates both parent and child report and then a final score is provided by the interviewer. The total score for the PARS is total of the 7 severity items. The total score ranges from 0 to 35. Higher numbers represent more anxiety symptoms therefore worse outcomes.
Time Frame: The PARS measure will be collected at the baseline appointment before subjects begin the cognitive training as well as after completing 8 cognitive training sessions in four weeks.
Population: We included all participants with pre and post PARS scores; due to incomplete/missing data, 7 participant scores were calculated for the cognitive training group, and 5 participant scores were calculated for the sham training group.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Cognitive Training Participants: Participants will complete 30-45 minute cognitive training program twice a week for four weeks.
  Cognitive Training Program: The cognitive training program has been designed by Dr. Sylvester. It is a simple computer game looking at some shapes and faces on a computer screen and pressing a button when a target shape appears.
  This is the first study to use this exact computer training regimen for testing in its ability to reduce symptoms of anxiety in children with anxiety disorders. Each session of the computer game takes approximately 45-60 minutes and subjects complete 8 total sessions over one month. The computer game involves paying attention to parts of the screen while distracting square boxes appear at other locations.
- Sham Training Participants: Participants to the assigned sham training did not have square box distractors appear. A target "X" appears at the location that participants are paying attention to and the subjects press a button when it appears.
Arm/Group | Cognitive Training Participants | Sham Training Participants
Number analyzed (Participants) | 7 | 5
units on a scale | -3.86 [-8.76 to 1.05] | -1.4 [-5.29 to 2.49]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other Adverse Events were not monitored/assessed as this novel treatment was a simple computer task with no risks.
Description: All-Cause Mortality, Serious, and Other Adverse Events were not monitored/assessed as the intervention was a simple computer task that children completed.
Groups:
- Sham Cognitive Training: Participants will complete 30-45 minute cognitive training program twice a week for four weeks.
  Cognitive Training Program: The cognitive training program has been designed by Dr. Sylvester. It is a simple computer game looking at some shapes and faces on a computer screen and pressing a button when a target shape appears.
  This is the first study to use this exact computer training regimen for testing in its ability to reduce symptoms of anxiety in children with anxiety disorders. Each session of the computer game takes approximately 45-60 minutes and subjects complete 8 total sessions over one month. The computer game involves paying attention to parts of the screen while distracting square boxes appear at other locations. A target "X" appears at the location that participants are paying attention to and the subjects press a button when it appears.
Arm/Group | Active Cognitive Training | Sham Cognitive Training
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
An important limitation of the present study is that there was no control group without any cognitive training and the sample size was small. Therefore, we cannot conclusively state that the task itself reduced anxiety as opposed to non-specific factors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT03790696/Prot_SAP_000.pdf